CLINICAL TRIAL: NCT03982251
Title: The Effects of Whole Body Vibration Training With Different Frequencies on Bone Health and Neuromotor Performance in Individuals With Chronic Stroke: A Randomized Controlled Trial.
Brief Title: The Effects of Whole Body Vibration in People With Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Marco Yiu-Chung Pang, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20140226001-03
Record Dates: First submitted 2019-06-06; First posted 2019-06-11 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Stroke
Keywords: vibration; bone; mucle; cerebrovascular accident; rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High frequency whole body vibration (Experimental): This group will receive a single 8-minute session of WBV therapy. The frequency of the vibration signals will be set at 30Hz.
  Interventions: Procedure: High frequency whole body vibration
- low frequency whole body vibration (Active Comparator): This group will receive a single 12-minute session of WBV. The frequency of the vibration signals will be set at 20 Hz.
  Interventions: Procedure: Low frequency whole body vibration

INTERVENTIONS:
Procedure: High frequency whole body vibration — 1 single session ( 8 minutes) of whole body vibration therapy at 30 Hz
  Other Names: Whole body vibration therapy (30Hz)
  Arms: High frequency whole body vibration
Procedure: Low frequency whole body vibration — 1 single session ( 12 minutes) of whole body vibration therapy at 20 Hz
  Other Names: Whole body vibration therapy (20Hz)
  Arms: low frequency whole body vibration

SUMMARY:
Whole body vibration (WBV) has been found to be useful in promoting bone health and muscle performance in older adults. To date, no study has examined the effects of different WBV frequencies on the properties of the muscle-bone unit in stroke patients. The overall aim of the proposed study is to compare the efficacy of different vibration frequencies on properties of the muscle function and bone turnover among people with chronic stroke.

It is hypothesized that the higher-vibration frequency protocol will lead to significantly better outcomes related to the bone turnover and muscle function.

DETAILED DESCRIPTION:
Whole body vibration (WBV) has been found to be useful in promoting bone health and muscle performance in older adults. To date, no study has examined the effects of different WBV frequencies on the properties of the muscle-bone unit in stroke patients. The overall aim of the proposed study is to compare the efficacy of different vibration frequencies on properties of the muscle function and bone turnover among people with chronic stroke.

It is hypothesized that the higher-vibration frequency protocol will lead to significantly better outcomes related to the bone turnover and muscle function in people with chronic stroke.

ELIGIBILITY:
Inclusion Criteria:

1. a diagnosis of stroke
2. stroke onset >6 months
3. >18 years of age
4. able to walk for short distance independently with or without walking aid
5. able to understand simple verbal commands

Exclusion Criteria:

1. neurological conditions other than stroke
2. significant musculoskeletal conditions (e.g. amputations)
3. metal implants in the lower extremity
4. previous fracture of the lower extremity
5. are currently taking bone resorption inhibitors or were taking the same before stroke.
6. significant peripheral vascular disease
7. vestibular disorders
8. pregnancy
9. Other serious illnesses that preclude the person from participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-08-28 (Actual)

PRIMARY OUTCOMES:
bone resorption marker | pre-test (week 0)
  Serum level of aminoterminal crosslinked telopeptide
bone resorption marker | post-test (week8)
  Serum level of aminoterminal crosslinked telopeptide

SECONDARY OUTCOMES:
Six Minute Walk Test | pre-test (week 0)
  endurance test
Six Minute Walk Test | post-test (week8)
  endurance Test
Gait velocity | pre-test (week 0)
  10-meter walking test
Gait velocity | post-test (week8)
  10-meter walking test
Spasticity | pre-test (week 0)
  H-reflex on tibial nerve and modified ashworth scale
Spasticity | post-test (week8)
  H-reflex on tibial nerve and modified ashworth scale

CONTACTS AND LOCATIONS:
Overall Officials: Marco YC Pang, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong